CLINICAL TRIAL: NCT04075513
Title: A 12-week Randomized, Controlled Trial to Compare TOUJEO® and TRESIBA® in Terms of Glucose Values in Target Range and Variability During Continuous Glucose Monitoring in Patients With Type 1 Diabetes Mellitus
Brief Title: Comparison of Glucose Values and Variability Between TOUJEO and TRESIBA During Continuous Glucose Monitoring in Type 1 Diabetes Patients
Acronym: inRange
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14947; 2017-002756-91 (EudraCT Number); U1111-1197-8171 (Other: UTN)
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Toujeo (Experimental): Toujeo (Insulin Glargine, 300 U/ml) subcutaneous (SC) injection, once daily in the morning before breakfast for 12 weeks on top of rapid acting insulin analog.
  Interventions: Drug: Insulin glargine, 300 U/ml; Drug: Background therapy: Rapid acting insulin analogs
- Tresiba (Active Comparator): Tresiba (Insulin Degludec, 100U/ml) SC injection, once daily in the morning before breakfast for 12 weeks on top of rapid acting insulin analog.
  Interventions: Drug: Insulin degludec, 100U/ml; Drug: Background therapy: Rapid acting insulin analogs

INTERVENTIONS:
Drug: Insulin glargine, 300 U/ml — Pharmaceutical form: solution for injection in a prefilled pen
  Route of administration: SC injection
  Other Names: Toujeo; HOE901-U300
  Arms: Toujeo
Drug: Insulin degludec, 100U/ml — Pharmaceutical form: solution for injection in a prefilled pen
  Route of administration: SC injection
  Other Names: Tresiba
  Arms: Tresiba
Drug: Background therapy: Rapid acting insulin analogs — Route of administration: SC injection

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of insulin glargine 300 units per milliliter (U/ml) in comparison to insulin degludec 100 U/ml on glycemic control and variability in participants with diabetes mellitus.

Secondary Objective:

To evaluate the glycemic control and variability parameters in each treatment group at Week 12 using Continuous Glucose Monitoring.

To evaluate the safety of insulin glargine 300 U/ml in comparison to insulin degludec 100 U/ml.

DETAILED DESCRIPTION:
The duration of the study per participant was around 18 weeks: 1 or 2 weeks of screening followed by a 4-week run-in period, a 12-week treatment period and a 2 to 4 days follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 1 Diabetes mellitus.
* Participants treated with multiple daily injections using basal insulin analog once daily and rapid acting insulin analogs for at least one year.
* HbA1c greater than or equal to (>=) 7 percent (%) (53 millimoles per mole [mmol/mol]) and less than or equal to (<=) 10% (86 mmol/mol) at screening.

Exclusion criteria:

* Participants not on stable dose of basal insulin analog.
* Participants having received Toujeo or Tresiba as basal insulin within 30 days prior to screening.
* Participants not having used the same insulins (both basal and rapid) within 30 days prior to screening.
* Participants having received basal insulin dose >= 0.6 units per kilogram body weight within 30 days prior to screening.
* Participants having received any glucose lowering drugs (including any premixed insulins, human regular insulin as mealtime insulins, any others injectable or oral), other than basal and rapid insulin analogs, within 3 months prior to screening.
* End stage renal disease or on renal replacement treatment.
* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months prior to screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Body weight change >=5 kilogram within 3 months prior to screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- United States, Dallas, Texas, United States
- Investigational site BRAZIL, Brazil, Brazil
- Investigational site Germany, Germany, Germany
- Investigational site Hungary, Hungary, Hungary
- Investigational site Netherlands, Netherlands, Netherlands
- Investigational site Turkey, Turkey, Turkey (Türkiye)
- Investigational site United Kingdom, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Battelino T, Bosnyak Z, Danne T, Mukherjee B, Edelman S, Pilorget V, Choudhary P, Renard E, Bergenstal R. InRange: Comparison of the Second-Generation Basal Insulin Analogues Glargine 300 U/mL and Degludec 100 U/mL in Persons with Type 1 Diabetes Using Continuous Glucose Monitoring-Study Design. Diabetes Ther. 2020 Apr;11(4):1017-1027. doi: 10.1007/s13300-020-00781-6. Epub 2020 Feb 25. PMID 32100192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 40 active sites in 7 countries. A total of 550 participants were screened between 09 October 2019 and 06 May 2021, of which 343 participants were enrolled and randomized by an interactive response technology (IRT) (1:1 ratio) to receive Toujeo or Tresiba. A total of 207 participants were screen failure mainly due to not meeting eligibility criteria.
Pre-assignment Details: Randomization was stratified by hemoglobin A1c (HbA1c) at screening (less than [<] 8.0 percent [%]; greater than or equal to [>=] 8.0%). Participants continued their short-acting mealtime insulin analogue (i.e., rapid insulin analogs) which they had used for at least 30 days before the screening visit and continued the same throughout the study.
Groups:
- Toujeo: Toujeo (Insulin Glargine, 300 units per milliliter [U/ml]) subcutaneous (SC) injection, once daily in the morning before breakfast for 12 weeks on top of rapid acting insulin analog.
- Tresiba: Tresiba (Insulin Degludec, 100 U/ml) SC injection, once daily in the morning before breakfast for 12 weeks on top of rapid acting insulin analog.
Period: Overall Study
Arm/Group | Toujeo | Tresiba
Started | 172 | 171
Completed | 164 | 167
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 4 | 2
Not completed — Switch to insulin pump | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population which included all randomized participants (who signed the informed consent form and were allocated to a treatment group before the first investigational medicinal product [IMP] administration and recorded in the IRT database), irrespective of the treatment actually received and were analyzed according to the treatment group allocated by randomization.
Groups:
- Toujeo: Toujeo (Insulin Glargine, 300 U/ml) SC injection, once daily in the morning before breakfast for 12 weeks on top of rapid acting insulin analog.
- Total: Total of all reporting groups
Arm/Group | Toujeo | Tresiba | Total
Number analyzed (Participants) | 172 | 171 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (13.53) | 42.8 (13.05) | 42.8 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 74 | 160
  Male | 86 | 97 | 183
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time of Glucose Concentration Within the Target Range of Greater Than or Equal to (>=) 70 to Less Than or Equal to (<=) 180 Milligrams Per Deciliter: Non-inferiority Analysis
Description: The Continuous Glucose Monitoring (CGM) system combined frequent interstitial glucose measurements (every 5 minutes) with ability to analyze glucose levels in real time. Adjusted least square (LS) means and standard error (SE) were obtained using analysis of covariance (ANCOVA) model on data obtained from the multiple imputations during Week 10 to Week 12.
Time Frame: During Week 10 up to Week 12
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of time | 52.74 (0.859) | 55.09 (0.893)
Statistical Analysis 1: Comparison: Toujeo vs Tresiba; Analysis was performed using ANCOVA model including the fixed categorical effect of treatment groups and randomization stratum of screening HbA1c (<8.0%, >=8.0%) and the continuous fixed covariate of Baseline percent time in range value; Test type: Non-Inferiority — Non-inferiority was based on a relative margin of 10%. Since higher time in range means better outcome, non-inferiority was demonstrated if the lower bound of the two-sided 95% confidence interval (CI) of the difference between Toujeo LS mean and 90% of Tresiba LS mean at Week 12 was > 0; p = 0.0067, ANCOVA — Threshold of significance at <0.05; Least square mean difference = 3.16, 95% CI 2-sided [0.88 to 5.44], Standard Error of Mean 1.163 — This estimation parameter corresponds to the difference between Toujeo LS mean and 90% of Tresiba LS mean

2. Secondary Outcome: Glucose Total Coefficient of Variation (CV%)
Description: CV% was a measure of spread of variability relative to mean of population. For CGM glucose values, CV% was measure of glycemic variability across 20 days and calculated as ratio of standard deviation of glucose values to mean of glucose values. LS means and SE were obtained using ANCOVA model using fixed categorical effects of treatment groups (Toujeo, Tresiba), randomization stratum of screening HbA1c (<8.0% versus >=8.0%), and the continuous fixed covariate of Baseline value.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total CV
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of total CV | 39.91 (0.360) | 41.22 (0.373)
Statistical Analysis 1: Comparison: Toujeo vs Tresiba; A hierarchical step-down testing procedure was used to control type I error. The hierarchical testing was then performed sequentially only when the primary endpoint demonstrated non-inferiority. Analysis was performed using ANCOVA model including the fixed categorical effect of treatment groups and randomization stratum of screening HbA1c (<8.0%, >=8.0%) and the continuous fixed covariate of Baseline percent time in range value; Test type: Non-Inferiority — Non-inferiority was based on a relative margin of 10%. Since lower CV means better outcome, non-inferiority was demonstrated if the upper bound of the two-sided 95% CI of the difference between Toujeo LS mean and 110% of Tresiba LS mean at Week 12 was < 0; p < 0.0001, ANCOVA — Threshold of significance at <0.05; Least square mean difference = -5.44, 95% CI 2-sided [-6.50 to -4.38], Standard Error of Mean 0.542 — This estimation parameter corresponds to the difference between Toujeo LS mean and 110% of Tresiba LS mean

3. Secondary Outcome: Percentage of Time of Glucose Concentration Within the Target Range of >=70 to <=180 Milligrams Per Deciliter: Superiority Analysis
Description: The CGM system combined frequent interstitial glucose measurements (every 5 minutes) with ability to analyze glucose levels in real time. Adjusted LS means and SE were obtained using ANCOVA model on data obtained from the multiple imputations during Week 10 to Week 12.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of time | 52.74 (0.859) | 55.09 (0.893)
Statistical Analysis 1: Comparison: Toujeo vs Tresiba; A hierarchical step-down testing procedure was used to control type I error. The hierarchical testing was then performed sequentially when the primary endpoint and the secondary endpoint of total CV demonstrated non-inferiority. Analysis was performed using ANCOVA model including the fixed categorical effect of treatment groups and randomization stratum of screening HbA1c (<8.0%, >=8.0%) and the continuous fixed covariate of Baseline percent time in range value; Test type: Superiority — Superiority was demonstrated if the lower bound of the two-sided 95% CI of the adjusted difference estimate of Toujeo and Tresiba at Week 12 was >0; p = 0.0548, ANCOVA — Threshold of significance at <0.05; Least square mean difference = -2.35, 95% CI 2-sided [-4.75 to 0.05], Standard Error of Mean 1.225

4. Secondary Outcome: Glucose Within-day CV% and Between-day CV%
Description: CV% was a measure of spread of variability relative to mean of population. For CGM glucose values, CV% was measure of glycemic variability across 20 days and calculated within day and between days as ratio of standard deviation of glucose values to mean of glucose values. LS mean and SE were obtained from ANCOVA model including fixed categorical effects of treatment groups (TOUJEO, TRESIBA), randomization stratum of screening HbA1c (<8.0% versus >=8.0%), and as well as, the continuous fixed covariate of Baseline value.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of CV
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of CV
  Within-day CV% | 33.48 (0.342) | 34.37 (0.351)
  Between-day CV% | 17.23 (0.404) | 18.08 (0.415)

5. Secondary Outcome: Change From Baseline in Glycated Hemoglobin A1c (HbA1c) at Week 12
Description: Change in HbA1c at Week 12 was analyzed using an ANCOVA model including the fixed categorical effects of treatment groups (Toujeo, Tresiba), and the continuous fixed covariate of Baseline HbA1c value.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 154 | 153
percentage of HbA1c | -0.75 (0.058) | -0.92 (0.057)

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: Change in FPG was analyzed using an ANCOVA model including the fixed categorical effects of treatment groups (Toujeo, Tresiba) and the randomization stratum of HbA1c at screening (<8.0%, >=8.0%) and the continuous fixed covariate of Baseline FPG value.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 154 | 151
milligrams per deciliter | -16.05 (5.455) | -34.55 (5.523)

7. Secondary Outcome: Percentage of Time With Glucose Level <70 Milligrams Per Deciliter (All Time and During the Night)
Description: The CGM system combined frequent interstitial glucose measurements (every 5 minutes) with ability to analyze glucose levels in real time. "All time" represent the time between 00.00 hour to 23.59 hours and "night" represent the time between 00.00 hour to 05.59 hours. LS means and SE were obtained using ANCOVA model using fixed categorical effects of treatment groups (Toujeo, Tresiba), randomization stratum of screening HbA1c (<8.0% versus >=8.0%), and the continuous fixed covariate of Baseline value.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of time
  All time | 5.55 (0.353) | 6.49 (0.362)
  Night | 6.32 (0.511) | 6.26 (0.524)

8. Secondary Outcome: Mean Hours Per Day With Glucose Level <70 Milligrams Per Deciliter (All Time and During the Night)
Description: "All time" represent the time between 00.00 hour to 23.59 hours and "night" represent the time between 00.00 hour to 05.59 hours. Mean hours per day with glucose level <70 milligrams per deciliter during "all time" and only "during night" for the duration of Week 10 to Week 12 is reported in this outcome measure.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
hours per day
  All time | 1.33 (0.085) | 1.56 (0.087)
  Night | 0.38 (0.031) | 0.38 (0.031)

9. Secondary Outcome: Percentage of Time With Glucose Level >180 Milligrams Per Deciliter
Description: The CGM system combined frequent interstitial glucose measurements (every 5 minutes) with ability to analyze glucose levels in real time. LS means and SE were obtained using ANCOVA model using fixed categorical effects of treatment groups (Toujeo, Tresiba), randomization stratum of screening HbA1c (<8.0% versus >=8.0%), and the continuous fixed covariate of Baseline value.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
percentage of time | 41.52 (0.975) | 38.31 (1.002)

10. Secondary Outcome: Mean Hours Per Day With Glucose Level >180 Milligrams Per Deciliter
Description: Mean hours per day with glucose level >180 milligrams per deciliter for the duration of Week 10 to Week 12 is reported in this outcome measure.
Time Frame: During Week 10 up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per day
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 158 | 151
hours per day | 9.96 (0.234) | 9.19 (0.240)

11. Secondary Outcome: Number of Participants With at Least One Hypoglycemic Event During the On-treatment Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because the participant was not capable of helping self. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <3.9 millimoles per liter (mmol/L) (<70 milligrams per deciliter). On-treatment period was defined as the time from the first injection of IMP (included) up to 2 days after the last injection of IMP.
Time Frame: From the first injection of IMP up to 2 days after the last injection of IMP (i.e., up to 86 days)
Population: Analysis was performed on safety population that included all randomized participants who had received at least one dose or part of a dose of IMP and were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 172 | 171
Participants
  Any hypoglycemia | 165 | 166
  Severe hypoglycemia | 8 | 10
  Documented symptomatic hypoglycemia | 136 | 134

12. Secondary Outcome: Number of Hypoglycemic Events Per Participant Year During the On-treatment Period
Description: Number of hypoglycemia events (any, severe and documented) per participant-year of exposure were reported. Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, because the participant was not capable of helping self. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <3.9 mmol/L (<70 milligrams per deciliter). On-treatment period was defined as the time from the first injection of IMP (included) up to 2 days after the last injection of IMP. Total participant years = The sum of the duration of exposure for all participants, expressed in participant years.
Time Frame: From the first injection of IMP up to 2 days after the last injection of IMP (i.e., up to 86 days)
Population: Analysis was performed on safety population.
Measure: Number; unit: events per participant-year
Arm/Group | Toujeo | Tresiba
Number analyzed (Participants) | 172 | 171
events per participant-year
  Any hypoglycemia | 109.4 | 114.9
  Severe hypoglycemia | 0.2 | 0.3
  Documented symptomatic hypoglycemia | 67.1 | 66.9

ADVERSE EVENTS:
Time Frame: From the first injection of IMP up to 2 days after the last injection of IMP (i.e., up to 86 days)
Description: Reported AEs were TEAEs that developed/worsened or became serious during on-treatment period (defined as the time from the first injection of IMP to the last injection of IMP + 2 days). Analysis was performed on safety population.
Groups:
- Toujeo: Toujeo (Insulin Glargine, 300 U/ml) SC injection, before meals once daily in the morning for 12 weeks on top of rapid acting insulin analog.
- Tresiba: Tresiba (Insulin Degludec, 100 U/ml) SC injection, before meals once daily in the morning for 12 weeks on top of rapid acting insulin analog.
Arm/Group | Toujeo | Tresiba
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/171
Serious Adverse Events (participants affected / at risk) | 7/172 | 8/171
Other Adverse Events (participants affected / at risk) | 0/172 | 0/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toujeo (N=172) | Tresiba (N=171)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoglycaemic Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 4 (4) | 2 (3)
Orthostatic Intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT04075513/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04075513/SAP_001.pdf